CLINICAL TRIAL: NCT01071629
Title: Aerobic Interval Training Versus Combined Aerobic Interval Training and Strength Training Effects in Patients With Heart Failure
Brief Title: Exercise Training Effects in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Serafim Nanas, MD, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOA-2010
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Heart Failure
Keywords: interval training; strength training; exercise capacity; chronic heart failure; Cardiac rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined interval and strength training (Active Comparator): CHF Pts randomly designed at the combined interval and strength training group
  Interventions: Other: Exercise training
- Aerobic interval training (Active Comparator): CHF Patients that randomly designed to participate at the interval training group
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Interval training (30 sec 50% of peak Work Rate achieved at the steep ramp test/60 sec recovery no exercise) for 40 min in the interval training group
  Arms: Aerobic interval training
Other: Exercise training — Interval training (30 sec 50% of peak Work Rate achieved at the steep ramp test/60 sec recovery no exercise) for 20 min and Strength training of the quadriceps, hamstrings, muscles of the shoulder and biceps brachialis for 20 min 3 times per week for 36 sessions
  Arms: Combined interval and strength training

SUMMARY:
Chronic heart failure (CHF) is a common syndrome characterized by several central hemodynamic and peripheral vascular and muscle abnormalities including autonomic imbalance, neuro-hormonal over-activation and decreased oxidative status.

In patients suffering from CHF, exercise confers several beneficial effects on the cardiovascular and peripheral systems, mainly by continuous aerobic training. However, interval aerobic training has also been validated as an alternate form of training that increases the exercise capacity of patients who are in CHF.

Recent studies have suggested that resistance training alone or as a complementary program besides the traditionally aerobic continuous training might exert favorable effects. However, little it is known about the combined effects of interval and strength training in CHF patients.

Aim of this prospective randomized controlled study was to investigate the effects of combined interval and strength training comparing to interval training alone in CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable systolic heart failure
* NYHA functional class ≤ III
* Optimal medical treatment

Exclusion Criteria:

* Contraindications for a maximal cardiopulmonary exercise testing (CPET) according to the American Thoracic Society/American College of Chest Physicians Statement
* Moderate to severe COPD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-11; Primary Completion 2010-04 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Aerobic exercise capacity | 3 months

SECONDARY OUTCOMES:
Endothelial function, oxygen kinetics, ventilatory drive | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Nanas, MD, Principal Investigator — University of Athens
Locations (1):
- Cardiopulmonary Exercise Testing & Rehabilitation Laboratory, First Critical Care Unit, School of Medicine, National & Kapodistrian University of Athens, Athens, Greece

REFERENCES:
- [Result] Anagnostakou V, Chatzimichail K, Dimopoulos S, Karatzanos E, Papazachou O, Tasoulis A, Anastasiou-Nana M, Roussos C, Nanas S. Effects of interval cycle training with or without strength training on vascular reactivity in heart failure patients. J Card Fail. 2011 Jul;17(7):585-91. doi: 10.1016/j.cardfail.2011.02.009. Epub 2011 Apr 22. PMID 21703531
- [Result] Tasoulis A, Papazachou O, Dimopoulos S, Gerovasili V, Karatzanos E, Kyprianou T, Drakos S, Anastasiou-Nana M, Roussos C, Nanas S. Effects of interval exercise training on respiratory drive in patients with chronic heart failure. Respir Med. 2010 Oct;104(10):1557-65. doi: 10.1016/j.rmed.2010.03.009. PMID 20663654
- [Result] Bouchla A, Karatzanos E, Dimopoulos S, Tasoulis A, Agapitou V, Diakos N, Tseliou E, Terrovitis J, Nanas S. The addition of strength training to aerobic interval training: effects on muscle strength and body composition in CHF patients. J Cardiopulm Rehabil Prev. 2011 Jan-Feb;31(1):47-51. doi: 10.1097/HCR.0b013e3181e174d7. PMID 20562711
- [Result] Gerovasili V, Drakos S, Kravari M, Malliaras K, Karatzanos E, Dimopoulos S, Tasoulis A, Anastasiou-Nana M, Roussos C, Nanas S. Physical exercise improves the peripheral microcirculation of patients with chronic heart failure. J Cardiopulm Rehabil Prev. 2009 Nov-Dec;29(6):385-91. doi: 10.1097/HCR.0b013e3181b4ca4e. PMID 19770806
- [Result] M.Kravari, I. Vasileiadis, V. Gerovasili, E. Karatzanos, A. Tasoulis, K. Kalligras, S. Drakos, S. Dimopoulos, M. Anastasiou-Nana, S. Nanas. Effects of a 3-month rehabilitation program on muscle oxygenation in congestive heart failure patients as assessed by NIRS. International Journal of Industrial Ergonomics 40(2): 212-217, 2010